CLINICAL TRIAL: NCT02264158
Title: A Double-blind, Randomised, Placebo Controlled, 6 Parallel Groups Study to Assess the Influence of Telmisartan (40 mg or 160 mg), Lacidipine (4 mg or 6 mg) and Their Combination (Telmisartan 40 mg and Lacidipine 4 mg) p.o. Once Daily for Seven Days on the QT Interval of the ECG in Healthy Male and Female Volunteers
Brief Title: Influence of Telmisartan and Lacidipine, Combined or Alone, on QT Interval in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.378
Record Dates: First submitted 2014-10-14; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy

ARMS (6):
- Telmisartan high (Experimental)
  Interventions: Drug: Telmisartan high
- Telmisartan low (Experimental)
  Interventions: Drug: Telmisartan low
- Lacidipine high (Active Comparator)
  Interventions: Drug: Lacidipine high
- Lacidipine low (Active Comparator)
  Interventions: Drug: Lacidipine low
- Telmisartan+Lacidipine (Experimental)
  Interventions: Drug: Telmisartan low; Drug: Lacidipine low
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan high
  Arms: Telmisartan high
Drug: Telmisartan low
  Arms: Telmisartan low; Telmisartan+Lacidipine
Drug: Lacidipine high
  Arms: Lacidipine high
Drug: Lacidipine low
  Arms: Lacidipine low; Telmisartan+Lacidipine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Assessment of the influence of telmisartan, lacidipine and their combination on the QTC interval of the ECG

ELIGIBILITY:
Inclusion Criteria:

All participants in the study should be healthy males/females, range from 21 to 50 years of age and their body mass index (BMI) be within 18.5 to 29.9 kg/m2.

In accordance with Good Clinical Practice and local legislation all volunteers will have given their written informed consent prior to admission to the study.

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, heart rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another tiral with an investigational drug (<= two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (>= 100 ml within four weeks prior to administration or during the trial)
* Any laboratory value outside the clinically accepted reference range
* Excessive physical activities within the last week before the trial or during the trial

Following exclusion criteria are of special interest for this study:

* Hypersensitivity to telmisartan, lacidipine and/or related drugs of these classes
* Supine blood pressure at screening of systolic <= 110 mmHg and diastolic <= 60 mmHg
* Any ECG value outside of the reference range of clinical relevance, but not limited to PR interval > 240 ms, QRS interval > 110 ms, QTcB > 470 ms for females and QTcB > 450 ms for males

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception (adequate contraception e.g. sterilisation, intrauterine pessary (IUP), oral contraceptives)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2001-09; Primary Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Average QTcF (QT interval Fridericia correction) change | baseline, day 1, day 7

SECONDARY OUTCOMES:
Change in QT interval | baseline, day 1, day 7
Change in QTcB (QT interval Bazett correction) interval | baseline, day 1, day 7
Change in PQ interval | baseline, day 1, day 7
Change in QRS interval | baseline, day 1, day 7
Change in RR interval | baseline, day 1, day 7
Change in heart rate (HR) | baseline, day 1, day 7
Occurrence of ECG abnormalities | baseline, day 1, day 7
Change in T wave morphology | baseline, day 1, day 7
  normal, flat, inverted, biphasic
Change in U wave morphology | baseline, day 1, day 7
  normal, abnormal
Area under the plasma concentration time curve (AUC) | day 1, day 7
Maximum plasma concentration (Cmax) | day 1, day 7
Time to attain maximum plasma concentration (tmax) | day 1, day 7
Trough plasma concentration at steady state (Cmin,ss) | day 7
Number of participants with adverse events | up to 8 days after last treatment